CLINICAL TRIAL: NCT07170046
Title: Predictive Value of CEA and ctDNA for Postoperative Recurrence in Patients With High CEA Sensitivity Lung Cancer
Brief Title: Predictive Value of CEA and ctDNA in Lung Cancer Recurrence
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2025-310
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-04

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort: The clinical information of the population in this cohort was retrospectively collected.
- prospective cohort: The clinical information of the population in this cohort was prospectively collected.

SUMMARY:
The study aims to investigate the predictive value of CEA levels for postoperative recurrence in the highly sensitive CEA lung cancer patients and to explore whether the dynamic changes of postoperative CEA and MRD in this population are related.This study was carried out to accurately predict the recurrence time, save the time and cost of changing the intervention strategy, and provide more personalized treatment for patients.

DETAILED DESCRIPTION:
This study will collect two groups of cohorts: prospective and retrospective.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative CEA > 5mg/l
2. MRD testing was conducted before the operation
3. The primary lesion was resected through surgery
4. There should be at least two CEA and MRD follow-up tests within 2 years after the operation
5. Postoperative pathology confirmed it as a malignant lung tumor

Exclusion Criteria:

1. Those without available imaging records
2. Patients with a history of malignant tumors within the past five years
3. Patients with secondary lung cancer

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Guangdong Provincial People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative tumor recurrence or progression | 2 years
  If the tumor recurs or progresses within 2 years, it will be marked as 1. If not, it will be marked as 0.

IPD SHARING:
Plan to Share IPD: Undecided